CLINICAL TRIAL: NCT04473443
Title: Addition of Computer Simulations to the Pre-procedural Planning to Minimize Adverse Events After Transcatheter Aortic Valve Implantation
Brief Title: Addition of Computer Simulations to Minimize Adverse Events After Transcatheter Aortic Valve Implantation
Acronym: PRECISE_TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Feops (Industry)
Responsible Party: Principal Investigator, Nicolas van Mieghem, principal investigator, Erasmus Medical Center
Other Study IDs: PRECISE TAVI
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Aortic Valve Stenosis; Bicuspid Cardiac Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients with a challenging anatomy, including bicuspid aortic valve, severely calcified aortic valves or small aortic roots
  Interventions: Other: FEops HEARTguideTM
- Cohort B: Consecutive patients eligible for TAVI with ACURATE-NEO2 valve
  Interventions: Other: FEops HEARTguideTM

INTERVENTIONS:
Other: FEops HEARTguideTM — A patient-specific computer simulation that aims to improve the outcomes after TAVI by suggesting THV platform, THV size and implantation depth with the use of the pre-procedural CT-scan.

SUMMARY:
The objective is to assess the influence of FEops HEARTguide on overall device success in TAVI patients with challenging anatomies (Cohort A) or in transcatheter heart valve (THV) platform selection (Cohort B).

DETAILED DESCRIPTION:
Rationale Transcatheter aortic valve implantation (TAVI) is increasingly used to treat patients with severe aortic stenosis. However, by extending the indication for TAVI, simulation may become increasingly important to improve procedure execution, safety and efficacy.

Objective Assess the influence of FEops HEARTguideTM on overall device success in challenging anatomies (Cohort A) or in transcatheter heart valve (THV) platform selection (Cohort B).

Study design Prospective, observational multi-center trial with 2 cohorts.

Study population

1. Cohort A: patients with challenging anatomy undergoing EvolutTM TAVI (Medtronic, Minneapolis, Minnesota), to evaluate the influence of FEops HeartGuideTM on overall device success through valve size and implantation depth.
2. Cohort B: consecutive patients, eligible for TAVI with ACURATE NEO2 TM (Boston Scientific, Marlborough, Massachusetts) to evaluate the influence of FEops heartGuideTM on overall device success and PVL prediction.

Main Endpoints

1. Overall device success conform VARC-2 including need for new permanent pacemaker. 2. Incidence of > trivial Paravalvular leakage (PVL) 3. Need for new permanent pacemaker

ELIGIBILITY:
Inclusion Criteria:

* Cohort A:

  1. Patients with a Bicuspid Aortic Valve (Sievers 0 or 1) or functional Bicuspid Aortic Valve
  2. Patients with a severely calcified aortic valve (Agatston score > 3000 for men, and > 1600 for women)
  3. Patients with small anatomy defined by mean aortic annulus diameter < 20mm
* Cohort B:

  1. every patient accepted for TAVI and eligible for ACURATE-NEO2-valve.

Exclusion Criteria:

* poor CT quality
* previous aortic valve replacement
* Permanent pacemaker at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective multi-center international Registry of TAVI patients include for Cohort A patients with the following complex anatomy: BAV (Sievers 0 or 1) or functional bicuspid aortic valves, severely calcified aortic valve and small aortic roots.
  And for Cohort B consecutive patients eligible for TAVI with ACURATE-NEO2-valve
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
overall device success conform the VARC-2 document | 30 days after TAVI
  * Incidence of mortality
  * incidence of stroke
  * incidence of major vascular complication
  * incidence of life-threatening bleeding

SECONDARY OUTCOMES:
incidence of more than trivial PVL | 30 days after TAVI
  total incidence of trivial PVL
conduction abnormalities and need for new permanent pacemaker implantation | 30 days after TAVI
  * incidence of new permanent pacemaker implantations
  * incidence of left bundle branch block
  * incidence of total AV block

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas van Mieghem, Md,PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. J Thorac Cardiovasc Surg. 2013 Jan;145(1):6-23. doi: 10.1016/j.jtcvs.2012.09.002. Epub 2012 Oct 16. PMID 23084102